CLINICAL TRIAL: NCT00914082
Title: The Effect of Mental Training on Childbirth Measured on Pain Experience and Other Birth Outcomes
Brief Title: Mental Training and Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-20080200
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Childbirth; Pain
Keywords: Self hypnosis; Hypnosis; mental training; antenatal training; pregnancy; pain control; Childbirth; Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- antenatal classes in self hypnosis (Experimental): 3 antenatal classes in self hypnosis. 3 audio compact discs for homework in self hypnosis and 1 audio compact disc for birth
  Interventions: Behavioral: Self hypnosis
- relaxation and awareness (Active Comparator): 3 antenatal classes including training in relaxation methods and mindfulness.3 audio compact discs for homework and 1 for birth.
  Interventions: Behavioral: Self hypnosis
- Control (Other): Only receive ordinary antenatal care and no additional interventions
  Interventions: Behavioral: Self hypnosis

INTERVENTIONS:
Behavioral: Self hypnosis — 3 antenatal classes of 1 hour. 3 audio compact discs for reenforcement. 1 audio compact discs for support at birth
  Other Names: Hypnosis

SUMMARY:
Labour pain is a challenge to the parturient woman. Pain relief methods during birth are limited and often associated with side effects. Several studies indicate that a mental trainings method, self hypnosis, has a positive impact on the labour pain and other birth outcomes.

The aim of this randomized controlled study is to examine the effect of a short antenatal course in self hypnosis on the use of epidural analgesia during birth and several other birth outcomes. Data collection includes questionnaires, register data, medical records and biological material.

DETAILED DESCRIPTION:
Background:

Experiencing labour pain is a challenge to the parturient woman and can possibly cause a traumatic birth experience, post traumatic stress syndrome, post partum depression, caesarean section or refraining from having more children.

Pharmacological pain relief methods to relieve birth pain are limited and often associated with side effects. Investigating new methods without adverse effects to relieve labour pain is therefore important.

Several studies indicate that a mental trainings method, self-hypnosis, has a positive impact on labour pain and several other birth outcomes. However, many of these studies were based on observational data with a limited amount of participants that may be prone to bias and confounding.

Aim:

The aim of this study is to examine the effect of a short antenatal course in self hypnosis on the use of epidural analgesia during childbirth.

Method:

The study is designed as an interventional single center study taking place at one of the largest birth departments in Denmark. It is a randomised, controlled, single blinded trial using a 3 arm group design.

The participants will be randomised by a voice respond program. The intervention group receives 3 antenatal classes in self hypnosis taught by midwives with qualified training in hypnosis. The course includes audio compact discs for homework in self hypnosis.

The active comparator group also receives 3 antenatal classes. The program is taught by the same midwives as in the intervention group and includes a mixture of training in different relaxation methods and mindfulness. This course also includes audio compact discs for homework.

The control group will only receive ordinary antenatal care and no additional interventions.

The data collection will be based on questionnaires, register data, medical records and biological material.

The endpoints are:

Primary:

* The use of epidural analgesia during birth

Secondary:

* Length of birth
* Birth progression at arrival at birth department
* Birth experience (pain, control, anxiety)
* Medical interventions during birth including mode of delivery
* Hemorrhage during birth
* Saliva cortisol profile at birth and 6 weeks p.p.
* Infection during birth and the first 6 weeks p.p. (mother and child)
* Postnatal depression
* Breastfeeding duration
* Child's condition and wellbeing at birth and 6 months later
* Future mode of delivery

At the start of the study, we performed our power calculations based on the fact that 44% of all primiparas at Aarhus University Hospital Skejby in 2007 had received epidural analgesia. We hypothesized that the observed frequency of epidural analgesia would be 25 % in the intervention group, 35 % in the placebo effect group and 40 % in the placebo group.

According to these power calculations, we should include 328 participants in the hypnosis group, 328 participants in the active comparator group and 152 participants in the control group to obtain a power of 80 % (α 0.05 (two sided)) in detecting a difference of 5 percentage points (relative risk (RR) 0.71) between the intervention and the active comparator group. By including 152 participants in the control group we would have a larger power to detect a difference of 15 percentage points (RR 0.63) in the use of epidural analgesia between the intervention and the control group.

Because we expected that some participants would develop medical conditions that required epidural analgesia during delivery, give birth prior to receiving their allocated intervention, or give birth by caesarean section, we decided to increase the sample size by 10% in all groups to a total of 890 participants.

In 2010, the study board experienced that in 2009 the general frequency of epidural analgesia in primiparas giving birth at Aarhus University Hospital Skejby had decreased to 34%.Therefore it was decided to adjust the sample size according to this new information.

When the sample size was adjusted we maintained the same sample ratios between the groups and hypothesized that the observed frequency of epidural analgesia would be 22 % in the intervention group, 30 % in the placebo effect group and 32 % in the placebo group. To obtain a power of 80 % (α 0.05 (two sided)) in detecting a difference of 8 percentage points (RR 0.73) between the intervention and the active comparator group in the use of epidural analgesia and a difference of 10 percentage points (RR 0.68) between the intervention and the control group we should include 446 participants in the hypnosis group, 446 participants in the active comparator group and 226 participants in the control group, in total 1097 participants. Again, we further increased the sample size with an extra 10% to account for those women that would not be able to comply with their allocated treatment because of obstetric conditions and reached a sample size in total of 1208.

Analyses will primarily be performed as "intended to treat". Secondary analyses according to "as treated" and preplanned subgroup analysis will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Nulliparous
* Planning a normal and vaginal birth

Exclusion Criteria:

* Poor understanding of Danish
* Psychological and psychiatric problems
* Medical disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1222 (Actual)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The use of epidural analgesia during birth | At birth

SECONDARY OUTCOMES:
Length of birth | At Birth
Birth progression at arrival at birth department | arrival at birth department
Birth experience (pain, control, anxiety) | 6 weeks p.p.
Medical interventions during birth including mode of delivery | At birth
Hemorrhage during birth | At birth
Saliva cortisol profile at birth and 6 weeks p.p. | at birth and 6 weeks p.p.
Infection during birth and the first 6 weeks p.p. (mother and child) | at birth and during the first 6 weeks p.p.
Postnatal depression | 6 weeks and 6 month p.p.
Breastfeeding duration | 6 weeks and 6 month p.p.
Childs condition and wellbeing at birth and 6 months later | At birth and 6 month p.p.
Future mode of delivery | 6 month p.p.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Werner, Ms of healthsc, Ph.Dstudent, Principal Investigator — Department of Gynecology and Obstetrics, Aarhus University Hospital Skejby; Niels Uldbjerg, MD, Professor, Study Chair — Department of Gynecology and Obstetrics, Aarhus University Hospital Skejby; Ellen A Nøhr, ass. professor, Study Chair — University of Aarhus, Department of Epidemiology; Bobby Zachariae, MD, Professor, Study Chair — Aarhus University Hospital, Psychooncology Research Unit; Aase M Hansen, senior researcher, Study Chair — National Research Center for the Working Enviroment
Locations (1):
- Department of Obstetrics and Gynecology, Aarhus University Hospital Skejby, Aarhus, Aarhus N, Denmark

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203
- [Derived] Werner A, Uldbjerg N, Zachariae R, Wu CS, Nohr EA. Antenatal hypnosis training and childbirth experience: a randomized controlled trial. Birth. 2013 Dec;40(4):272-80. doi: 10.1111/birt.12071. PMID 24344708
- [Derived] Werner A, Uldbjerg N, Zachariae R, Nohr EA. Effect of self-hypnosis on duration of labor and maternal and neonatal outcomes: a randomized controlled trial. Acta Obstet Gynecol Scand. 2013 Jul;92(7):816-23. doi: 10.1111/aogs.12141. Epub 2013 Apr 22. PMID 23550694
- [Derived] Werner A, Uldbjerg N, Zachariae R, Rosen G, Nohr EA. Self-hypnosis for coping with labour pain: a randomised controlled trial. BJOG. 2013 Feb;120(3):346-53. doi: 10.1111/1471-0528.12087. Epub 2012 Nov 27. PMID 23190251